CLINICAL TRIAL: NCT00006111
Title: Multicenter Study of the Quality of Life of Patients With Invasive Urothelial Cancer Treated With Conservative Surgery Followed by Cisplatin, Fluorouracil and Radiotherapy
Brief Title: Surgery Plus Combination Chemotherapy and Radiation Therapy in Treating Patients With Cancer of the Urinary Tract
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068123; FRE-FNCLCC-97015; EU-20009
Record Dates: First submitted 2000-08-03; First posted 2004-02-03 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bladder Cancer; Transitional Cell Cancer of the Renal Pelvis and Ureter; Urethral Cancer
Keywords: stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; anterior urethral cancer; posterior urethral cancer; urethral cancer associated with invasive bladder cancer; metastatic transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter
MeSH Terms: conditions — Urinary Bladder Neoplasms; Urethral Neoplasms | interventions — Cisplatin; Fluorouracil; Radiotherapy

ARMS (2):
- resectable disease (Experimental)
  Interventions: Drug: cisplatin; Drug: fluorouracil; Procedure: conventional surgery; Radiation: radiation therapy
- unresectable disease (Experimental)
  Interventions: Drug: cisplatin; Drug: fluorouracil; Radiation: radiation therapy

INTERVENTIONS:
Drug: cisplatin
Drug: fluorouracil
Procedure: conventional surgery
  Arms: resectable disease
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining surgery with chemotherapy and radiation therapy may be an effective way to treat cancer of the urinary tract.

PURPOSE: Phase II trial to study the effectiveness of combining surgery, chemotherapy and radiation therapy in treating patients who have stage II, stage III, or stage IV cancer of the urinary tract .

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the quality of life of patients with invasive stage II, III, or IV carcinoma of the urothelium treated with conservative surgery plus cisplatin, fluorouracil, and radiotherapy. II. Determine the efficacy of this regimen, in terms of local control, in these patients. III. Determine survival of patients treated with this regimen. IV. Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to tumor type (T2-4a, N0, M0; potentially resectable; no contraindication to surgery vs T2-4b, N0 or N1 or pN1, M0; refused surgery or medical contraindications to surgery). (Accrual for stratum I was completed as of 10/23/2001.) Stratum I (resectable disease): Regimen A: Patients undergo radiotherapy 5 days a week for 5 weeks. Patients also receive fluorouracil IV continuously and cisplatin IV continuously on days 1-4 during weeks 1 and 4. If complete response is achieved by week 5, patients proceed to regimen B. If partial response or progression is observed, patients undergo cystectomy. If cystectomy is refused, patients proceed to regimen B. Regimen B: Patients undergo radiotherapy 5 days a week for 2 weeks. Patients also receive fluorouracil and cisplatin as in regimen A on weeks 2 and 5. (Accrual for stratum I was completed as of 10/23/2001.) Stratum II (unresectable disease): Patients undergo radiotherapy 5 days a week for 7 weeks. Patients also receive fluorouracil and cisplatin as in regimen A on weeks 1, 4, and 7. Quality of life is assessed at baseline, at 6 months, and then at 1 year. Patients are followed at 6-8 weeks, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 75 patients (35 for stratum I and 40 for stratum II) will be accrued for this study. (Accrual for stratum I was completed as of 10/23/2001.)

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage II, III, or IV carcinoma of the urothelium infiltrating muscle Primary OR After development of a superficial tumor T2-T4b with or without lymph node involvement and no detectable metastases No epidermoid cancer or adenocarcinoma No extrapelvic lymph node involvement

PATIENT CHARACTERISTICS: Age: 18 to 70 Performance status: WHO 0-2 Life expectancy: More than 6 months Hematopoietic: WBC greater than 4,000/mm3 Platelet count greater than 100,000/mm3 Neutrophil count greater than 1,500/mm3 Hemoglobin greater than 10 g/dL Hepatic: Not specified Renal: Creatinine less than 1.5 mg/dL Other: Not pregnant Fertile patients must use effective contraception during and for 2 months after study No other prior malignancy except nonmelanomatous skin cancer or carcinoma in situ of the cervix No prior serious illness of the gastrointestinal tract (e.g., rectal bleeding or diverticulosis with complications) No contraindication to fluorouracil, cisplatin, or radiotherapy

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy except intravesicular instillations Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy Surgery: Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 1999-04 (Actual); Primary Completion 2003-01 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Leon Lagrange, MD, Study Chair — Centre Antoine Lacassagne
Locations (11):
- France (11):
  - Institut Sainte Catherine, Avignon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - C.H.U. - Hopital Gaston Doumergue, Nîmes
  - Centre Eugene Marquis, Rennes
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Hospitalier General de Saint Nazaire, Saint-Nazaire
  - Institut Claudius Regaud, Toulouse
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy